CLINICAL TRIAL: NCT04638374
Title: Adaptation of Lumbar Spine to a Mattress: a MRI Evaluation.
Acronym: Mattress&Spine
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Other Study IDs: Mattress & Spine
Record Dates: First submitted 2020-11-16; First posted 2020-11-20 (Actual); Last update posted 2020-11-30 (Actual); Status verified 2020-11

CONDITIONS: Lumbar Spine Adaptation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
People spend almost a third of their life sleeping and understanding how the spine can adapt to a mattress is essential for promoting people's health. The general objective of this study is to study and evaluate the adaptation of the spine to a mattress. The primary objective is the assessment of the variation in the lumbar lordosis angle (sagittal plane) in the supine position, on a mattress, compared to the value measured in the supine position on a rigid surface.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 45 years old
* Female or Male sex
* Cognitive integrity
* Absence of usual contraindications to MRI

Exclusion Criteria:

* Clinical condition diagnosed by a doctor
* Spinal pathologies
* Pregnant woman
* Claustrophobia

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy people between 18 and 45 years of age.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2020-11-04 (Actual); Primary Completion 2021-08-31 (Estimated); Study Completion 2021-10-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of lumbar section of spine in a supine position on a mattress | 10 minutes
  Magnetic Risonance is used to assess the spine
Evaluation of lumbar section of spine in a supine position without mattress | 10 minutes
  Magnetic Risonance is used to assess the spine

SECONDARY OUTCOMES:
Evaluation of lumbar section of spine in a standing position | 2 minutes
  EOS is used to assess the spine

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Istituto Ortopedico Galeazzi, Milan, Italy

REFERENCES:
- [Derived] Vitale JA, Borghi S, Bassani T, Messina C, Sconfienza LM, Galbusera F. Effect of a mattress on lumbar spine alignment in supine position in healthy subjects: an MRI study. Eur Radiol Exp. 2023 Sep 4;7(1):47. doi: 10.1186/s41747-023-00361-w. PMID 37661237